CLINICAL TRIAL: NCT04619290
Title: Treatment in Outpatient Patients With Covid-19 With Methylene Blue and Photodynamic
Brief Title: Outpatient Treatment With CoVid-19 With Prexablu
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Reg. Lic. Adolfo Lopez Mateos (Other Government)
Responsible Party: Principal Investigator, M. Eunice Rodríguez Arellano, Principal Investigator, Hospital Reg. Lic. Adolfo Lopez Mateos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 064.I.2020
Record Dates: First submitted 2020-11-04; First posted 2020-11-06 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Sars Cov 2
Keywords: COVID-19; methylene blue; photodynamic interval therapy; outpatient; Mexico
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Single group comparison with contemporaneous conventionally treated patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene blue treated group (Experimental): Patients will be included in this group with the following symptoms: with at least one of the following symptoms: headache, nausea, dyspnea, myalgia, vomiting. Also that they meet the inclusion criteria
  Interventions: Drug: Sublingual Methylene blue
- Conventionally treated group (Active Comparator): Patients will be included in this group with the following symptoms: with at least one of the following symptoms: headache, nausea, dyspnea, myalgia, vomiting. Also that they meet the inclusion criteria
  Interventions: Other: Control patients

INTERVENTIONS:
Drug: Sublingual Methylene blue — Patients will be received the treatment as follow: it will be placed Low Level Light Therapy (LLLT) NocUlite on the ventral side of the wrist on full power. Draw out 1ml of diluted Prexablu into a syringe. Activate this syringe LLLT device for 10 minutes. Then place 1ml of this activated solution of Prexablu sublingually. Patients must keep the solution under the tongue for 10 minutes before swallowing. Keep wrist pads on patients for 50 minutes.
  Arms: Methylene blue treated group
Other: Control patients — Control patients will be received the conventional treatment that may include analgesic, anti-inflammatory, antibiotic, steroid, antiplatelet, and anticoagulant.
  Arms: Conventionally treated group

SUMMARY:
Within the epidemic context of phase 3 in Mexico, the implementation of new treatments that have been shown to be beneficial for patients in other countries is an urgent need. Methylene blue (MB, the oxidized form, blue color) has been used in many different clinical medicine areas, ranging from malaria to orthopedics. Methylene blue absorbs energy directly from a light source and then transfers this energy to molecules of oxygen creating singlet oxygen (O2), which is the first electronic excited state of molecular oxygen (O2). Singlet oxygen is extremely electrophilic; thus, it can directly oxidize electron-rich double bonds in biological molecules and macromolecules. For this reason, methylene blue has been used as a photosensitizer in the treatment of cancer and the protection of serum from viral agents. Methylene blue can be reactivated using energy from a light source in the body until processed out through the kidneys.

DETAILED DESCRIPTION:
Patients diagnosed with COVID-19 and confirmed positive with the virus by PCR will be treated with Prexablu for seven days. The administration is Sublingual 1 ml Prexablu once a day and PDT for 1 hour daily x 7 days. Days to clinical improvement to be evaluated for seven days considering temperature and other vital signs measurement, arterial oxygen saturation.

I. On day one and day seven a blood sample will be drawn to assess chemistry (including liver function tests), C reactive protein, IgG, IgM, IL-6, erythrocyte sedimentation rates like procalcitonin, ferritin levels, and the D dimer II. Daily PCR Swabs measuring cycle threshold (CT) will be collected (days 1 - 7) III. Daily 1ml Prexablu will be placed sublingual

1. Prexablu activated for 10 minutes with Low Level Light Therapy (670 nm light) before being placed sublingually.
2. Low Level Light Therapy (NocUlite device) will be placed on wrist for 50 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Of both sexes
* Confirmed case of Covid-19 (by RT-PCR) and CT less than 32 in the E
* That they go to the ER service due to COVID symptoms, and that they voluntarily agree to participate in the study by written the informed consent
* With at least 1 of the following symptoms: fever, headache, nausea, dyspnea, myalgia, vomiting, or diarrhea
* With chest X-ray without pneumonia criteria
* With SO2> 90
* No history of allergic reaction to methylene blue
* No history of treatment with medication with methylene blue negative interaction

Exclusion Criteria:

* Pregnancy and breastfeeding
* Preadmission anticoagulation
* Severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2)
* Active chronic hepatitis
* Patients with history of allergic reaction or significant sensitivity to methylene blue
* Treatment with immunosuppressive agents
* Diagnosis of cancer at any stage and of any type.
* Pregnancy and breastfeeding
* Patients who plan to become pregnant during the study period or within 6 months after the end of the study period.
* Participation in another clinical trial with an experimental drug in the last 30 days.
* Other pathologies that, in the medical opinion, contraindicate participation in the study.
* Uncompensated comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change form baseline in Arterial oxygen saturation | up to 7 days
  Aretrial oxygen saturation will be taken by an oximeter
Days to clinical improvement | up to 7 days
  Number of days of patient discharge

SECONDARY OUTCOMES:
Change Form Baseline in C reactive protein at 7 days | up to 7 days
  Blood samples will be taken on days 1 and 7
Change Form Baseline in IL-1β | up to 7 days
  Blood samples to analyse IL-1β will be taken on days 1 and 7.
Change Form Baseline in Erythrocyte sedimentation rate like procalcitonin | up to 7 days
  Blood samples to analyse the Erythrocyte sedimentation rate like procalcitonin
Change Form Baseline in Ferritin levels | up to 7 days
  Blood samples to analyse Ferritin levels
Change Form Baseline in D dimer | up to 7 days
  Blood samples to analyse D dimer will be taken on days 1 and 7

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Lic Adolfo Lopez Mateos, Mexico City, Ciudad de Mexico CDMX (Mexico City), Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Ji W, Wang W, Zhao X, Zai J, Li X. Cross-species transmission of the newly identified coronavirus 2019-nCoV. J Med Virol. 2020 Apr;92(4):433-440. doi: 10.1002/jmv.25682. PMID 31967321
- [Background] Baud D, Qi X, Nielsen-Saines K, Musso D, Pomar L, Favre G. Real estimates of mortality following COVID-19 infection. Lancet Infect Dis. 2020 Jul;20(7):773. doi: 10.1016/S1473-3099(20)30195-X. Epub 2020 Mar 12. No abstract available. PMID 32171390
- [Background] Backer JA, Klinkenberg D, Wallinga J. Incubation period of 2019 novel coronavirus (2019-nCoV) infections among travellers from Wuhan, China, 20-28 January 2020. Euro Surveill. 2020 Feb;25(5):2000062. doi: 10.2807/1560-7917.ES.2020.25.5.2000062. PMID 32046819
- [Background] Wang W, Xu Y, Gao R, Lu R, Han K, Wu G, Tan W. Detection of SARS-CoV-2 in Different Types of Clinical Specimens. JAMA. 2020 May 12;323(18):1843-1844. doi: 10.1001/jama.2020.3786. PMID 32159775
- [Background] Oz M, Lorke DE, Hasan M, Petroianu GA. Cellular and molecular actions of Methylene Blue in the nervous system. Med Res Rev. 2011 Jan;31(1):93-117. doi: 10.1002/med.20177. PMID 19760660
- [Background] Bradberry SM. Occupational methaemoglobinaemia. Mechanisms of production, features, diagnosis and management including the use of methylene blue. Toxicol Rev. 2003;22(1):13-27. doi: 10.2165/00139709-200322010-00003. PMID 14579544
- [Background] Barbosa P, Peters TM. The effects of vital dyes on living organisms with special reference to methylene blue and neutral red. Histochem J. 1971 Jan;3(1):71-93. doi: 10.1007/BF01686508. No abstract available. PMID 4106597
- [Background] Wainwright M, Crossley KB. Methylene Blue--a therapeutic dye for all seasons? J Chemother. 2002 Oct;14(5):431-43. doi: 10.1179/joc.2002.14.5.431. PMID 12462423
- [Background] Lee SK, Mills A. Novel photochemistry of leuco-Methylene Blue. Chem Commun (Camb). 2003 Sep 21;(18):2366-7. doi: 10.1039/b307228b. PMID 14518917
- [Background] Khan S, Alam F, Azam A, Khan AU. Gold nanoparticles enhance methylene blue-induced photodynamic therapy: a novel therapeutic approach to inhibit Candida albicans biofilm. Int J Nanomedicine. 2012;7:3245-57. doi: 10.2147/IJN.S31219. Epub 2012 Jun 29. PMID 22802686
- [Background] Wainwright M. Methylene blue derivatives--suitable photoantimicrobials for blood product disinfection? Int J Antimicrob Agents. 2000 Dec;16(4):381-94. doi: 10.1016/s0924-8579(00)00207-7. PMID 11118846
- [Background] Tardivo JP, Del Giglio A, de Oliveira CS, Gabrielli DS, Junqueira HC, Tada DB, Severino D, de Fatima Turchiello R, Baptista MS. Methylene blue in photodynamic therapy: From basic mechanisms to clinical applications. Photodiagnosis Photodyn Ther. 2005 Sep;2(3):175-91. doi: 10.1016/S1572-1000(05)00097-9. Epub 2005 Nov 21. PMID 25048768
- [Background] Tuite EM, Kelly JM. Photochemical interactions of methylene blue and analogues with DNA and other biological substrates. J Photochem Photobiol B. 1993 Dec;21(2-3):103-24. doi: 10.1016/1011-1344(93)80173-7. PMID 8301408
- [Background] Eickmann M, Gravemann U, Handke W, Tolksdorf F, Reichenberg S, Muller TH, Seltsam A. Inactivation of Ebola virus and Middle East respiratory syndrome coronavirus in platelet concentrates and plasma by ultraviolet C light and methylene blue plus visible light, respectively. Transfusion. 2018 Sep;58(9):2202-2207. doi: 10.1111/trf.14652. Epub 2018 May 6. PMID 29732571
- [Background] Chatterjee GC, Noltmann EA. Dye-sensitized photooxidation as a tool for the elucidation of critical amino acid residues in phosphoglucose isomerase. Eur J Biochem. 1967 Jul;2(1):9-18. doi: 10.1111/j.1432-1033.1967.tb00098.x. No abstract available. PMID 6079766
- [Background] Triesscheijn M, Baas P, Schellens JH, Stewart FA. Photodynamic therapy in oncology. Oncologist. 2006 Oct;11(9):1034-44. doi: 10.1634/theoncologist.11-9-1034. PMID 17030646
- [Background] Faddy HM, Fryk JJ, Hall RA, Young PR, Reichenberg S, Tolksdorf F, Sumian C, Gravemann U, Seltsam A, Marks DC. Inactivation of yellow fever virus in plasma after treatment with methylene blue and visible light and in platelet concentrates following treatment with ultraviolet C light. Transfusion. 2019 Jul;59(7):2223-2227. doi: 10.1111/trf.15332. Epub 2019 May 3. PMID 31050821
- [Background] Fryk JJ, Marks DC, Hobson-Peters J, Watterson D, Hall RA, Young PR, Reichenberg S, Tolksdorf F, Sumian C, Gravemann U, Seltsam A, Faddy HM. Reduction of Zika virus infectivity in platelet concentrates after treatment with ultraviolet C light and in plasma after treatment with methylene blue and visible light. Transfusion. 2017 Nov;57(11):2677-2682. doi: 10.1111/trf.14256. Epub 2017 Jul 17. PMID 28718518
- [Background] Eickmann M, Gravemann U, Handke W, Tolksdorf F, Reichenberg S, Muller TH, Seltsam A. Inactivation of three emerging viruses - severe acute respiratory syndrome coronavirus, Crimean-Congo haemorrhagic fever virus and Nipah virus - in platelet concentrates by ultraviolet C light and in plasma by methylene blue plus visible light. Vox Sang. 2020 Apr;115(3):146-151. doi: 10.1111/vox.12888. Epub 2020 Jan 12. PMID 31930543
- [Background] Ziv G, Heavner JE. Permeability of the blood-milk barrier to methylene blue in cows and goats. J Vet Pharmacol Ther. 1984 Mar;7(1):55-9. doi: 10.1111/j.1365-2885.1984.tb00879.x. PMID 6708167
- [Background] Albert M, Lessin MS, Gilchrist BF. Methylene blue: dangerous dye for neonates. J Pediatr Surg. 2003 Aug;38(8):1244-5. doi: 10.1016/s0022-3468(03)00278-1. PMID 12891503
- [Background] Sills MR, Zinkham WH. Methylene blue-induced Heinz body hemolytic anemia. Arch Pediatr Adolesc Med. 1994 Mar;148(3):306-10. doi: 10.1001/archpedi.1994.02170030076017. PMID 8130867
- [Background] McFadyen I. The dangers of intra-amniotic methylene blue. Br J Obstet Gynaecol. 1992 Feb;99(2):89-90. doi: 10.1111/j.1471-0528.1992.tb14458.x. No abstract available. PMID 1554680
- [Background] Dolk H. Methylene blue and atresia or stenosis of ileum and jejunum. EUROCAT Working Group. Lancet. 1991 Oct 19;338(8773):1021-2. doi: 10.1016/0140-6736(91)91885-x. No abstract available. PMID 1681328
- [Background] van der Pol JG, Wolf H, Boer K, Treffers PE, Leschot NJ, Hey HA, Vos A. Jejunal atresia related to the use of methylene blue in genetic amniocentesis in twins. Br J Obstet Gynaecol. 1992 Feb;99(2):141-3. doi: 10.1111/j.1471-0528.1992.tb14473.x. PMID 1554667
- [Background] Iyengar B, Lal SK. Methylene blue and organised differentiation in the chick embryo. Acta Anat (Basel). 1985;123(4):220-3. doi: 10.1159/000146005. PMID 4061041
- [Background] Tiboni GM, Lamonaca D. Transplacental exposure to methylene blue initiates teratogenesis in the mouse: preliminary evidence for a mechanistic implication of cyclic GMP pathway disruption. Teratology. 2001 Oct;64(4):213-20. doi: 10.1002/tera.1066. PMID 11598927